CLINICAL TRIAL: NCT01970228
Title: Prospective Intra-individual Comparison of 18F-FDG and 68Ga-citrate PET/CT in Symptomatic Total Hip Arthroplasty Patients
Brief Title: Imaging of Joint Replacement Complications by PET/CT
Acronym: Propeli
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: T125/2012; EVO13086 (Other: Turku University Hospital)
Record Dates: First submitted 2013-09-19; First posted 2013-10-28 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Adverse Reactions to Metal Debris; Infection of Total Hip Joint Prosthesis; Mechanical Loosening of Prosthetic Joint

STUDY DESIGN:
Intervention Model Description: Intra-individual comparison of two diagnostic PET imaging tracers
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adverse reaction to metal debris (Active Comparator): 68Ga-citrate and 19F-FDG PET/CT imaging of hip replacement patients with adverse tissue reactions to metal debris
  Interventions: Diagnostic Test: 68Ga-citrate and 18F-FDG PET/CT imaging
- Periprosthetic joint infection (Active Comparator): 68Ga-citrate and 19F-FDG PET/CT imaging of hip replacement patients with periprosthetic joint infection
  Interventions: Diagnostic Test: 68Ga-citrate and 18F-FDG PET/CT imaging
- Aseptic mechanical implant loosening (Active Comparator): 68Ga-citrate and 19F-FDG PET/CT imaging of patients with aseptic mechanical loosening of hip prosthesis
  Interventions: Diagnostic Test: 68Ga-citrate and 18F-FDG PET/CT imaging

INTERVENTIONS:
Diagnostic Test: 68Ga-citrate and 18F-FDG PET/CT imaging — Single-day study of the two PET tracers

SUMMARY:
Total hip replacement is the well-established surgical method for treatment of hip osteoarthritis and related diseases. The outcome of the procedure is commonly satisfactory and most patients will not need any revision surgery. However, the procedure has its complications, including (1) periprosthetic infection, (2) mechanical loosening caused by wear particles and (3) adverse reaction caused by metal ions released from metal-on-metal bearing surfaces. The unsolved clinical problem is related to the differential diagnosis of these conditions. The purpose of this prospective clinical study is to compare the efficacy of two techniques of PET/CT imaging in the differential diagnosis of these complications. Positron Emission Tomography (PET)/Computed Tomography (CT) imaging, performed during a single day, will include the head-to-head comparison of 18F-Fluoro-D-Glucose (18F-FDG) PET/CT and 68Gallium-citrate (68Ga-citrate) PET/CT imaging.

DETAILED DESCRIPTION:
(68Ga) gallium citrate is a novel PET tracer aimed for detection of skeletal infections. It has not been previously applied to diagnose periprosthetic joint infections in arthroplasty patients. This exploratory prospective study, representing the first of its kind, examines the use of 68Ga-citrate as a diagnostic tool of periprosthetic infections aside with 18F-FDG tracer as the standard reference.

The first study group (n=10) will include total hip replacement patients without infection. The recruited patients should suffer from pain and/or functional impairment due to adverse reaction to metal debris (ARMD) caused by metal-on-metal bearings. The diagnosis of ARMD should be based on metal artifact reduction sequence magnetic resonance imaging (MARS-MRI). The patients will undergo the same-day comparison of the two PET/CT tracers.

The second study group (n=10) will include total hip replacement patients with bacteriologically confirmed periprosthetic joint infection. The third group (n=10) will include patients with aseptic loosening of total hip prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with uncemented total hip replacement
* American Society of Anesthesiology score I-III
* Group 1: local symptoms and MRI findings of the operated hip fulfilling the criteria of ARMD due to metal-on-metal bearings of the hip prosthesis, infection ruled out
* Group 2: bacteriologically verified periprosthetic infection of the hip prosthesis
* Group 3: local symptoms and radiographic findings of the hip prosthesis fulfilling the criteria of aseptic mechanical implant loosening, infection ruled out

Exclusion Criteria:

* any related condition of the index hip which requires immediate surgical intervention, such as a septic infection or a periprosthetic fracture
* any systemic disorder or condition (ASA IV) which makes the patient an unlikely candidate for revision surgery of the affected hip implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Exclusion of the presence of periprosthetic joint infection in ARMD patients | Clinical follow-up of 3 years or more after PET/CT imaging
  The two PET imaging techniques are expected to rule out infection in patients with ARMD due to metal-on-metal bearings

CONTACTS AND LOCATIONS:
Overall Officials: Hannu T Aro, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Background] Lankinen P, Lehtimaki K, Hakanen AJ, Roivainen A, Aro HT. A comparative 18F-FDG PET/CT imaging of experimental Staphylococcus aureus osteomyelitis and Staphylococcus epidermidis foreign-body-associated infection in the rabbit tibia. EJNMMI Res. 2012 Jul 23;2(1):41. doi: 10.1186/2191-219X-2-41. PMID 22824200
- [Background] Lankinen P, Makinen TJ, Poyhonen TA, Virsu P, Salomaki S, Hakanen AJ, Jalkanen S, Aro HT, Roivainen A. (68)Ga-DOTAVAP-P1 PET imaging capable of demonstrating the phase of inflammation in healing bones and the progress of infection in osteomyelitic bones. Eur J Nucl Med Mol Imaging. 2008 Feb;35(2):352-64. doi: 10.1007/s00259-007-0637-5. Epub 2007 Nov 24. PMID 18038133
- [Background] Makinen TJ, Lankinen P, Poyhonen T, Jalava J, Aro HT, Roivainen A. Comparison of 18F-FDG and 68Ga PET imaging in the assessment of experimental osteomyelitis due to Staphylococcus aureus. Eur J Nucl Med Mol Imaging. 2005 Nov;32(11):1259-68. doi: 10.1007/s00259-005-1841-9. Epub 2005 Jul 9. PMID 16007423
- [Background] Koort JK, Makinen TJ, Knuuti J, Jalava J, Aro HT. Comparative 18F-FDG PET of experimental Staphylococcus aureus osteomyelitis and normal bone healing. J Nucl Med. 2004 Aug;45(8):1406-11. PMID 15299068
- [Background] Ahtinen H, Kulkova J, Lindholm L, Eerola E, Hakanen AJ, Moritz N, Soderstrom M, Saanijoki T, Jalkanen S, Roivainen A, Aro HT. (68)Ga-DOTA-Siglec-9 PET/CT imaging of peri-implant tissue responses and staphylococcal infections. EJNMMI Res. 2014 Aug 8;4:45. doi: 10.1186/s13550-014-0045-3. eCollection 2014. PMID 25520903